CLINICAL TRIAL: NCT00961038
Title: Randomized, Single-Blinded, Placebo-Controlled Study to Evaluate the Safety and Tolerability, the Pulmonary Deposition and Pharmacokinetics of Ciprofloxacin in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (GOLD II - III), Following Inhalation of Ciprofloxacin PulmoSphere® Inhalation Powder
Brief Title: Study to Evaluate the Safety and Pharmacokinetics of Inhaled Ciprofloxacin in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 13014; 2008-006771-79 (EudraCT Number)
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2014-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Ciprofloxacin; Inhalation; Pharmacokinetics; Safety; Tolerability; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration | interventions — Ciprofloxacin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Ciprofloxacin (PulmoSphere, BAYQ3939)
- Arm 2 (Experimental)
  Interventions: Drug: Ciprofloxacin (PulmoSphere, BAYQ3939)
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciprofloxacin (PulmoSphere, BAYQ3939) — 32.5 mg ciprofloxacin betaine corresponding to 50 mg Ciprofloxacin PulmoSphere inhalation powder will be given as an initial single-dose inhalation (day 0).During the multiple-dose phase (day 2 to day 11), the same dose will be given twice daily, with a concluding single dose (on day 12)
  Arms: Arm 1
Drug: Ciprofloxacin (PulmoSphere, BAYQ3939) — 48,75 mg ciprofloxacin betaine corresponding to 75 mg Ciprofloxacin PulmoSphere inhalation powder will be given as an initial single-dose inhalation (day 0).During the multiple-dose phase (day 2 to day 11), the same dose will be given twice daily, with a concluding single dose (on day 12)
  Arms: Arm 2
Drug: Placebo — Placebo inhalation powder will be given as an initial single-dose inhalation (day 0).During the multiple-dose phase (day 2 to day 11), placebo will be given twice daily, with a concluding single dose (on day 12)
  Arms: Arm 3

SUMMARY:
Objectives of the study are to investigate the safety, tolerability and levels of ciprofloxacin in the lung after single and multiple inhalative administration to patients with moderate to severe COPD (stage II-III according to GOLD Criteria)

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with COPD, 40 to 75 years of age
* Diagnosis of COPD
* Airway obstruction with a post-bronchodilator Forced Expiratory Volume (FEV1) of >/=30% and </=65% of predicted and a post-bronchodilator FEV1 / Forced Vital Capacity (FVC) of </=70%
* Current or ex-smokers with a smoking history of more than 10 pack-years
* Patients must be able to produce acceptable induced sputum samples (as defined in the Study Procedure Manual)
* Normal body weight: Body Mass Index (BMI) between 19 and 35 kg/m2

Exclusion Criteria:

* Significant respiratory disease other than COPD as bronchial asthma, Cystic fibrosis or clinically evident bronchiectasis
* More than one COPD exacerbation within 12 months and within 8 weeks prior to screening
* total blood eosinophil count >/=600/mm3
* Thoracotomy with pulmonary resection
* Regularly use of daytime oxygen therapy for more than one hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy during clinic visits
* Hypersensitivity to the investigational drug or to other quinolones and/or to inactive constituents of the inhalation powder
* Hypersensitivity of the bronchial system to inhalation of nebulized drugs or saline solution
* Patients with a history of severe allergies, non-allergic drug reactions, or multiple drug allergies
* Concomitant use of medication which could interfere with the investigational drug. Before study drug administration a wash out period of more than 5 half lives has to be considered
* Concomitant inhalative therapy with antibiotics and/or concomitant systemic therapy with

  * fluoroquinolones
  * Oral beta-andrenergics, beta blockers
  * oral steroids
  * Methylxanthines: 24-hour washout of short-acting theophylline and 48-hour washout of long-acting theophylline prior to pre-study examination
  * Antihistamines, antileukotrienes prescribed for asthma
  * oral cromolyn sodium or oral nedocromil sodium

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Vital signs | Within 28 days after first treatment
Electrocardiogram (ECG) | Within 28 days after first treatment
Pulmonary function test | Within 28 days after first treatment
Pulse-oximetry | Within 12 days after first treatment

SECONDARY OUTCOMES:
Ciprofloxacin concentrations in blood | Within 14 days after first treatment
Ciprofloxacin concentrations in urine | Within 14 days after first treatment
Ciprofloxacin concentrations in sputum | Within 14 days after first treatment
Ciprofloxacin concentrations in mouth fluid | Within 7 days after first treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Hanover, Lower Saxony, Germany